CLINICAL TRIAL: NCT03112148
Title: A Phase 1, Randomized, Open Label, Partial Crossover Study To Evaluate The Pharmacokinetics And Safety Of Three Age-appropriate Modified Release Formulations And The Immediate Release Solution Of Tofacitinib In Healthy Adult Volunteers
Brief Title: PK Study in Adult Healthy Volunteers to Assess QD Dosing With the Selected Age-appropriate MR Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A3921261
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment A (Experimental): Single oral 10 mg dose of tofacitinib MR-FAST administered in the fed state.
  Interventions: Drug: 10 mg dose MR formulations,10 mg dose of tofacitinib IR solution
- Treatment B: (Experimental): Single oral 10 mg dose of tofacitinib MR-SLOW administered in the fed state.
  Interventions: Drug: 10 mg dose MR formulations,10 mg dose of tofacitinib IR solution
- Treatment C (Experimental): Single oral 10 mg dose of tofacitinib MR-FAST administered in the fasted state.
  Interventions: Drug: 10 mg dose MR formulations,10 mg dose of tofacitinib IR solution
- Treatment D (Experimental): Single oral 10 mg dose of tofacitinib MR-SLOW administered in the fasted state.
  Interventions: Drug: 10 mg dose MR formulations,10 mg dose of tofacitinib IR solution
- Treatment E (Experimental): Single oral 10 mg dose of tofacitinib MR-MODERATE administered in the fasted state
  Interventions: Drug: 10 mg dose MR formulations,10 mg dose of tofacitinib IR solution
- Treatment F (Experimental): Single oral 10 mg dose of tofacitinib IR Solution (10 mL of the 1 mg/mL solution) administered in the fasted state
  Interventions: Drug: 10 mg dose MR formulations,10 mg dose of tofacitinib IR solution

INTERVENTIONS:
Drug: 10 mg dose MR formulations,10 mg dose of tofacitinib IR solution — For the the relative bioavailability (BA) assessment , the investigational product(s) are:
  Test: 10 mg dose of age-appropriate MR formulations (MR-fast, MR-moderate, MR-slow). Each formulation contains 0.025 mg of tofacitinib/mg of microsphere. Reference: 10 mg dose of tofacitinib IR solution (1 mg of tofacitinib/mL).
  For the the food effect assessment, the investigational product(s) are:
  Test: 10 mg dose of age-appropriate MR formulations (MR-fast or MR-slow) c-oadministered with high-fat FDA breakfast. Reference: 10 mg dose of age-appropriate MR formulations (MR-fast or MR-slow) administered under fasted state.

SUMMARY:
This is a Phase 1, randomized, open label, 4-period, 6-sequence, partial cross-over, single-dose study to evaluate the PK of age-appropriate tofacitinib MR formulations (release rates: MR-Slow, MR-Moderate, and MR-Fast) compared to tofacitinib IR solution under fasting conditions. The effect of food on the PK of MR-Slow and MR-Fast will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive.
* Female subjects of nonchildbearing potential must meet at least 1 of the following criteria:

  1. Achieved postmenopausal status, defined as: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state;
  2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
  3. Have medically confirmed ovarian failure. All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 kg per m2; and a total body weight above 50 kg (110 lbs) for males and above 45 kg (99 lbs) for females.
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Clinically significant infections within the past 3 months, evidence of any infection within the past 7 days, history of disseminated herpes simplex infection or recurrent (>1 episode) herpes zoster or disseminated herpes zoster.
* Absolute lymphocyte count at Screening or Baseline less than the lower limit of the reference range for the local laboratory
* Evidence or history of cyclic neutropenia.
* Personal or family history of hereditary immunodeficiency
* Vaccination with live or attenuated vaccines within the 6 weeks of dosing, or is to be vaccinated with these vaccines at any time during study treatment or within 6 weeks following discontinuation of dosing.
* Any condition possibly affecting drug absorption (eg, gastrectomy, colon resection, etc.).
* History of, or current positive results for any of the following serological tests: human immunodeficiency virus (HIV), hepatitis B, or hepatitis C;
* Malignancy or a history of malignancy, with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
* Positive urine drug test.
* History of regular alcohol consumption
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement ) or 5 half-lives preceding the first dose of investigational product (whichever is longer).
* Nursing females or females of childbearing potential. Male subjects who are unwilling or unable to use a condom plus a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.

Herbal supplements and hormone replacement therapy must be discontinued at least 28 days prior to the first dose of investigational product.

* Use of CYP3A4 inhibitors or inducers within 14 days or 5 half-lives (whichever is longer) prior to dosing.
* Consumption of grapefruit or grapefruit-related citrus fruits (eg, Seville oranges, pomelos) or juices within 7 days prior to dosing.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] (AUCinf ) | 0.5, 1, 2, 3, 4, 5, 6, 9, 21, 24, 36, and 48 hours post dose
  Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0.5, 1, 2, 3, 4, 5, 6, 9, 21, 24, 36, and 48 hours post dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) of Modified Release (MR) formulation compared to Immediate Release (IR) solution
Maximum Observed Plasma Concentration (Cmax) | predose, 0.5, 1, 2, 3, 4, 5, 6, 9, 21, 24, 36, and 48 hours post dose
  Maximum (or peak) plasma concentration of MR formulation compared to IR solution
Time to Reach Maximum Observed Plasma Concentration (Tmax) | predose, 0.5, 1, 2, 3, 4, 5, 6, 9, 21, 24, 36, and 48 hours post dose
  Maximum time to peak plasma concentration of MR formulation compared to IR solution

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921261&StudyName=A+Phase+1%2C+Randomized%2C+Open+Label%2C+Partial+Crossover+Study+To+Evaluate+The+Pharmacokinetics+And+Safety+Of+Three+Age-appropriate+Modified+Release+Formulations+And+The+Immediate+Release+Solution+Of+Tofacitinib+In+Healthy+Adult+Volunteers